CLINICAL TRIAL: NCT03593551
Title: Investigation of Different Relaxation Interventions on Physical and Psychological Changes in Breastfeeding Mothers in China: A Pilot Study
Brief Title: Effects of Different Relaxation Interventions on Reducing Stress in Chinese Breastfeeding Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Principal Investigator, Mary Fewtrell, Professor of Paediatric Nutrition, University College, London
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 12681/001
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Stress-related Problem; Breastfeeding; Relaxation Therapy; Psychological Stress
Keywords: stress; anxiety; breastfeeding; relaxation; meditation; music
MeSH Terms: conditions — Breast Feeding; Stress, Psychological; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: within study design
Masking Description: The order for five treatments and one control are randomly allocated to participants. Each participant will attend all six sessions (five treatments and one control)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- relaxation and control (Experimental): All participants will attend five relaxation treatments and one control. The order of treatments and control will be randomised allocated to participants.
  Interventions: Combination Product: five relaxation treatments and one control

INTERVENTIONS:
Combination Product: five relaxation treatments and one control — Five treatments are relaxation meditation tape, music tape, relaxation lighting, meditation tape plus lighting, and music plus lighting. The control session have no intervention, participants will just be asked to sit comfortably for 10 minutes.

SUMMARY:
This pilot study aims to find the most effective relaxation technique to help primiparous mothers who are breastfeeding their infant. The effect of five different relaxation techniques on physical and psychological changes in Chinese mothers will be investigated. The interventions to be used in this study include: guided relaxation meditation tape, music tape, relaxation lighting, combined relaxation meditation and lighting, and combined music and lighting.

DETAILED DESCRIPTION:
The study will be conducted at Beijing Children Hospital, Beijing, China. A within-subject design will be used to evaluate the effectiveness and participants' feeling towards the five tested interventions compared to a control situation.

Population and recruitment The study population will be breastfeeding women in China. Recruitment will be take place through social media and community flyers in Beijing Children Hospital. Advertisements will be posted in the hospital while flyers will be sent to local communities. Interested women can make contact by email. Details about the study will be explained in the information sheet. After checking the eligibility and obtaining written informed consent, all eligible participants will be enrolled in the study.

Sample size calculation

To estimate the sample size of this pilot study, standard formulas used for calculation are:

Sample size (per equal-sized group) =8 x standard deviation ÷ (difference) 2

Here the effect size and standard deviation (SD) are estimated from a previous research, which evaluated the effect of audio-visual imagery on patient anxiety and physiological parameters. A sample of 51 patients was able to demonstrate a significant reduction in HR (mean change (Z)= -0.75, SD= 1.00; p=0.01). Accordingly, the estimated sample size (per equal-sized group) would be 28. However, since the present study will use a within-subject design, a sample of 14 participants will likely be able to demonstrate changes. Considering the potential drop-out rates, a total of 15-20 subjects will be enrolled in this study.

Study Procedures After obtaining informed consent, all participants enrolled in this study will be asked to attend for 30 minutes once to three times per week for five relaxation treatments and one control treatment (no intervention). The emotions and feelings of participants in both intervention and control treatment will be assessed before and after each treatment or control.

The duration of this study is six weeks. In order to fit with the subject's schedule and control the circadian rhythm, all treatments and control sessions will take place on different days each week. Each participant can choose a 30-minute time slot to fit participants' timetable. To make the outcome assessment more consistent, participants are encouraged to come at the same time of the day they chose. The order of interventions will be randomly assigned for each participant. Both relaxation interventions and control will be conducted in the breastfeeding room located at Beijing Children Hospital. This room is private, quiet and has comfy seating. Participants will be asked to leave their personal belongings, including any electronic devices, books and magazines, and personal work, during the experiment period.

Outcome measurements Primary outcomes of this study will be perceived relaxation level. Secondary outcomes are heart rate (HR), blood pressure (BP) and fingertip temperature (FT).

The HR, BP and FT will be measured at both the start and the end of the experiment. An automatic BP machine will be used for the measurements of HR and BP. The BP will be measured three times and the mean of three will be calculated and recorded. A thermometer will be used for the FT measurement.

The perceived relaxation will be assessed by a visual analogue scale (VAS), which consists of a horizontal 10cm line with one end representing the maximum and the other end the minimum of the variable to be measured. The right anchor of the scale is labelled as "completely relaxed" and the left anchor as "completely unrelaxed". Participants indicate their state of relaxation by marking a point along the line before each session and again at the end of each session. The distance from the left anchor to the mark made by participants is measured in millimeters and pre and post-test differences are compared.

Statistical analysis Data will be analysed using SPSS 24.0. Paired t-test will be used to detect changes in each of the primary outcomes before and after the treatment. One-way ANOVA will be conducted to find differences between control and each intervention group. Post-hoc analysis will be used to compare the effectiveness of each treatment. Differences will be considered statistically significant at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* primiparous mothers who are currently breastfeeding their infants
* generally healthy (without any diseases that could influence their blood pressure, heart rate, energy expenditure, or breastfeeding practice)
* did not attend any other intervention studies within 12 months

Exclusion Criteria:

* Smoker

Ages: 23 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological sex is female (breastfeeding mothers)
Enrollment: 20 (Actual)
Dates: Start 2018-06-03 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Perceived relaxation | 3 minutes
  Perceived relaxation measured by a visual analogue scale which consists of a horizontal 10cm line.The right anchor of the scale is identified as "completely relaxed" and the left anchor as"completely unrelaxed".

SECONDARY OUTCOMES:
Fingertip temperature | 10 seconds
  Fingertip temperature measured by Digital Body Thermometer in degrees centigrade. (A higher temperature is an indication of greater relaxation).
Heart rate | 2 minutes
  Heart rate measured by electronic blood pressure machine. A lower heart rate indicates greater relaxation.
Blood pressure | 2 minutes
  Systolic and diastolic pressure measured by electronic blood pressure machine. A lower BP indicates greater relaxation.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Fewtrell, PhD, Principal Investigator — University College, London
Locations (1):
- Beijing Children Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT03593551/Prot_001.pdf